CLINICAL TRIAL: NCT03395171
Title: Vitamin D3 Supplementation and Stress Fracture Occurrence in High-Risk Collegiate Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048420
Record Dates: First submitted 2017-12-22; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Vitamin D Deficiency; Stress Fracture; Athletic Injuries; Orthopedic Disorder
MeSH Terms: conditions — Vitamin D Deficiency; Fractures, Stress; Athletic Injuries; Musculoskeletal Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Cholecalciferol (Vitamin D3) (Experimental): Athletes with Vitamin D levels lower than 30ng/mL will be treated with the supplement for eight weeks.
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3)
- Prospective Control Group (No Intervention): Athletes with Vitamin D levels higher than 30ng/mL were enrolled and compared but not treated.

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vitamin D3) — Supplementation of subjects who meet the inclusion criteria and test to have below the threshold of vitamin D in their blood.
  Arms: Treatment: Cholecalciferol (Vitamin D3)

SUMMARY:
The main objective of this study is to find a correlation between vitamin D deficiency and stress fracture occurrences in athletes who participate in high-risk activities. These high-risk athletes undergo elevated bone turnover, which requires adequate levels of vitamin D in order to support bone health. It is hypothesized that providing supplemental treatment to athletes showing lower than normal serum vitamin D levels will decrease the occurrence of stress fractures. By recording the dates and specific occurrences of fractures, it may be possible to correlate injury rates with seasons, providing more supportive data to pre-existing literature.

This area of research is lacking in the quantity of prospective studies. Previous studies primarily focus on adolescent, elder, or military recruit populations. While literature has shown that vitamin D plays an important role in bone health, there are no previous studies that directly examine vitamin D deficiency and supplemental treatment in conditioned collegiate athlete populations. This study will add to the existing knowledge and will provide a more specific analysis for athletes.

DETAILED DESCRIPTION:
This study will focus on athletes who are at a higher risk of lower extremity stress fractures. Specifically, this study will be looking at male and female athletes on the track, cross-country, soccer, and basketball teams at the University of South Carolina. During the pre-season physical of each student athlete, serum vitamin D levels will be taken and recorded. There will be a certified nurse to draw the blood samples. This will take place at the University of South Carolina Athletic Department and/or the Palmetto Health Lab at 2 Medical Park. Potentially, every athlete of the given teams will be enrolled in the study unless they choose not to. Only subjects showing concentrations below 30 ng/mL, which is indicative of insufficient or deficient levels, will be provided supplemental treatment of 25-(OH) vitamin D. Every enrolled subject will be monitored for injury throughout the season. Any and all injuries will be positively identified, and any confirmed stress fractures will be recorded. Data from prospective seasons will be compared to an incidence percentage of athletes from previous seasons. Previous athletes did not receive any vitamin D treatment. These will be used as a control to determine if treatment affected the occurrence of stress fractures. All physicals and tests will be performed at the University of South Carolina Sports Medicine clinic by the sports medicine staff.

ELIGIBILITY:
Inclusion Criteria:

* Athlete on one of the following teams at local University: Men/Women Track and Field, Soccer, Basketball, and Women's Cross Country.

Exclusion Criteria:

* Athlete currently diagnosed with a stress fracture
* Athlete recovering from a lower extremity musculoskeletal injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence and prevalence of stress fractures in athlete cohorts | 5 Years
  To compare the incidence and prevalence of student athletes experiencing stress fractures during the 2015-16 academic year with the five previous years of reported data.

CONTACTS AND LOCATIONS:
Overall Officials: J. Benjamin Jackson III, MD, Principal Investigator — Prisma Health-Midlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03395171/Prot_SAP_000.pdf